CLINICAL TRIAL: NCT00631917
Title: A 54 Week, Randomized, Double-blind, Parallel-group, Multicenter Study Evaluating the Long-term Gastrointestinal (GI) Safety and Tolerability of Aliskiren (300 mg) Compared to Ramipril (10 mg) in Patients With Essential Hypertension
Brief Title: A Study Evaluating the Gastrointestinal (GI) Safety and Tolerability of Aliskiren Compared to Ramipril in Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Study Director, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100A2404
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, ramipril, colonoscopy
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental): For the first 2 weeks of the study, participants received aliskiren 150 mg once a day and were then forced titrated to aliskiren 300 mg once a day for 52 weeks. Participants also received a placebo capsule to match ramipril once a day for the study duration.
  Interventions: Drug: Aliskiren; Other: Placebo to Ramipril
- Ramipril (Active Comparator): For the first 2 weeks of the study participants received 5 mg ramipril orally once a day and were then forced titrated to ramipril 10 mg once a day for 52 weeks. Participants also received placebo to aliskiren for the duration of the study.
  Interventions: Drug: Ramipril; Other: Placebo to Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg once a day
  Arms: Aliskiren
Drug: Ramipril — Ramipril 10 mg once a day
  Arms: Ramipril
Other: Placebo to Ramipril — Placebo capsules to match ramipril.
  Arms: Aliskiren
Other: Placebo to Aliskiren — Placebo tablets to match aliskiren.
  Arms: Ramipril

SUMMARY:
This study will evaluate the long-term gastrointestinal (GI) safety and efficacy of aliskiren (300 mg) compared to ramipril (10mg) in patients ≥ 50 years with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, 50 years of age and older with a diagnosis of essential hypertension
* Successful high quality colonoscopy at baseline including visualization of the entire colon and the cecum as confirmed by a photograph and collection of the rectal and cecal mucosal biopsy samples
* All rectal, colon or cecal polyps found at baseline colonoscopy must be completely resected endoscopically at the time of the procedure.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation have been clearly explained to them (written informed consent).

Exclusion Criteria:

* Previously treated in an aliskiren study.
* Current evidence of inflammatory bowel disease, the presence of colonic ulcerations (or other indices of colitis of any type) or colorectal carcinoma including carcinoma in situ found at baseline colonoscopy.
* History of gastrointestinal carcinoma, Crohn's disease, ulcerative colitis, microscopic colitis.
* History of familial polyposis or hereditary nonpolyposis colorectal cancer.
* History of confirmed diverticulitis within 12 months of Visit 1.
* History of celiac disease (gluten intolerance).
* History of or current evidence on the baseline colonoscopy of melanosis coli.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — 862-778-8300
Locations (7):
- Investigative Site, Kansas City, Missouri, United States
- Investigative Site, Investigative Site, Argentina
- Investigative Site, Investigative Site, Colombia, Colombia
- Investigative Site, Investigative Site, France
- Investigative Site, Investigative Site, Germany
- Investigative Site, Investigative Site, India
- Investigative Site, Investigative Site, Spain

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren | Ramipril
Started | 375 | 399
Completed | 287 | 291
Not Completed | 88 | 108
Not completed — Adverse Event | 34 | 45
Not completed — Abnormal laboratory value(s) | 2 | 1
Not completed — Abnormal test procedure result(s) | 3 | 2
Not completed — Unsatisfactory therapeutic effect | 8 | 14
Not completed — No longer required study drug | 0 | 1
Not completed — Protocol deviation | 6 | 5
Not completed — Subject withdrew consent | 25 | 33
Not completed — Lost to Follow-up | 7 | 7
Not completed — Administrative problems | 2 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Ramipril | Total
Number analyzed (Participants) | 375 | 399 | 774
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (6.99) | 59.3 (6.65) | 59.3 (6.81)
Age, Customized [Number; unit: Participants]
  < 65 years | 299 | 313 | 612
  65 years and greater | 76 | 86 | 162
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 194 | 388
  Male | 181 | 205 | 386

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Colonic Pathology
Description: The primary analysis variable was the occurrence of an abnormal colonoscopy finding (defined as hyper-plastic polyps, inflammatory polyps, adenomatous polyps or carcinoma) at or prior to the planned one year visit. The occurrence of colonic pathology was identified during colonoscopy and histopathologic examination of biopsy. The composite endpoint was evaluated after one year of treatment with an aliskiren-based regimen compared to a ramipril-based regimen.
Time Frame: 54 weeks
Population: Primary Analysis Set, consisting of all randomized patients that had post-baseline colonoscopy procedure performed.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren | Ramipril
Number analyzed (Participants) | 314 | 325
Percentage of participants | 25.5 | 25.1

2. Secondary Outcome: Percentage of Participants With Each of the Individual Components of Colonic Pathology
Description: Assessment of the occurrence of the individual components (hyperplastic polyps, inflammatory polyps, adenomatous polyps or carcinomas) of the composite endpoint (colonic pathology) following one-year of treatment with an aliskiren-based regimen compared to a ramipril-based regimen.
Time Frame: 54 weeks
Population: Primary analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren | Ramipril
Number analyzed (Participants) | 314 | 325
Percentage of Participants
  Hyperplastic polyps | 13.1 | 10.2
  Inflammatory polyps | 0.0 | 0.3
  Adenomatous polyps | 15.0 | 17.3
  Carcinoma | 0.0 | 0.0

3. Secondary Outcome: Mucosal Hyperplasia Score in Rectal and Cecal Mucosal Biopsy Specimens After One Year of Treatment
Description: Maximum hyperplasia score at end of study across rectal and cecal mucosa biopsy specimens. Score of 0 is no change from baseline, the minimum possible score. Score > 0 is worsening from baseline in which the maximum possible score is 3.
Time Frame: 54 weeks
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Aliskiren | Ramipril
Number analyzed (Participants) | 314 | 325
participants
  Score = 0 | 295 | 304
  Score = 1 | 17 | 19
  Score = 2 | 0 | 0
  Score = 3 | 0 | 0
  Score is Missing | 2 | 2

4. Secondary Outcome: Percentage of Participants Achieving the Mean Sitting Blood Pressure Control Target
Description: The mean sitting blood pressure control target is defined as less than 140/90 mmHg (or 130/80 mmHg for diabetic patients)
Time Frame: Weeks 8, 30 and End of Study (54 weeks)
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren | Ramipril
Number analyzed (Participants) | 374 | 394
Percentage of Participants
  Week 8 | 50.8 | 44.9
  Week 30 | 60.2 | 54.1
  End of Study | 65.0 | 56.1

5. Primary Outcome: Summary of the End of Study Colonoscopy Results
Description: During each colonoscopy procedure, random biopsy samples were taken from normal appearing mucosa in both the cecum and rectum in addition to obvious endoscopically atypical areas. The mucosal biopsy samples were evaluated for mucosal hyperplasia, dysplasia, and inflammation. Anything noted as a distinct visual abnormality from cecum to rectum such as ulcers, erythematous mucosa, or polyps, was photographed and biopsied for histopathology evaluation. Colonic lesions were categorized according to location in the colon, size, number, and morphology.
Time Frame: 54 weeks
Population: Primary Analysis Set, consisting of all randomized patients that had post-baseline colonoscopy procedure performed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren | Ramipril
Number analyzed (Participants) | 314 | 325
Percentage of Participants
  Complete colonoscopy performed | 100 | 100
  Was cecum reached in procedure | 99.7 | 100
  Photos obtained | 99.4 | 99.7
  Took drug affecting bowel function | 0.0 | 0.6
  Took low dose aspirin during wk prior to procedure | 4.8 | 5.2
  Adequacy of bowel preparation - Optimal | 72.3 | 73.5
  Adequacy of bowel preparation - Suboptimal | 27.4 | 25.5
  Adequacy of bowel preparation - Inadequate | 0.3 | 0.9
  Colonoscopy prep given- PEG containing solution | 96.8 | 97.2
  Colonoscopy prep given - Other | 3.2 | 2.8
  Occurrence of colon polyps | 29.6 | 26.5
  Patients with polyps-Cecum/ascending | 11.8 | 11.4
  Patients with polyps-Transverse | 6.1 | 5.2
  Patients with polyps-Descending/sigmoid | 12.1 | 11.7
  Patients with polyps-Rectum | 8.0 | 6.5
  Mean number of polyps-Cecum/ascending | 1.3 | 1.2
  Mean number of polyps-Transverse | 1.2 | 1.4
  Mean number of polyps-Descending/sigmoid | 1.5 | 1.5
  Mean number of polyps-Rectum | 1.6 | 1.3
  Polyps were completely resected-Cecum/ascending | 11.8 | 11.1
  Polyps were completely resected-Transverse | 6.1 | 4.9
  Polyps were completely resected-Descending/sigmoid | 12.1 | 11.7
  Polyps were completely resected-Rectum | 7.6 | 6.5
  Photo taken for polyps-Cecum/ascending | 11.8 | 11.1
  Photo taken for polyps-Transverse | 5.7 | 4.6
  Photo taken for polyps-Descending/sigmoid | 10.8 | 10.5
  Photo taken for polyps-Rectum | 7.6 | 6.2
  Mucosal abnormalities for colitis | 1.3 | 1.5
  Patients with colitis-Cecum/ascending | 0.6 | 0.9
  Patients with colitis-Transverse | 0.0 | 0.0
  Patients with colitis-Descending/sigmoid | 0.0 | 0.0
  Patients with colitis-Rectum | 0.6 | 0.6
  Area of colitis biopsied-Cecum/ascending | 0.6 | 0.9
  Area of colitis biopsied-Transverse | 0.0 | 0.0
  Area of colitis biopsied-Descending/sigmoid | 0.0 | 0.0
  Area of colitis biopsied-Rectum | 0.6 | 0.6
  Area of colitis photographed-Cecum/ascending | 0.6 | 0.9
  Area of colitis photographed-Transverse | 0.0 | 0.0
  Area of colitis photographed-Descending/sigmoid | 0.0 | 0.0
  Area of colitis photographed-Rectum | 0.6 | 0.6
  Normal mucosal biopsies collected-Cecum | 99.4 | 99.7
  Normal mucosal biopsies collected-Rectum | 99.7 | 99.7
  Mean number of normal mucosal biopsies-Cecum | 3.0 | 3.0
  Mean number of normal mucosal biopsies-Rectum | 3.0 | 3.0
  Malignance for any biopsy samples-Yes | 0.0 | 0.0
  Malignance for any biopsy samples-No | 99.4 | 98.8
  Malignance for any biopsy samples-Missing | 0.6 | 0.9
  Inflammation for any biopsy samples-Yes | 1.0 | 0.6
  Inflammation for any biopsy samples-No | 98.4 | 98.8
  Inflammation for any biopsy samples-Missing | 0.6 | 0.6

ADVERSE EVENTS:
Arm/Group | Aliskiren | Ramipril
Serious Adverse Events (participants affected / at risk) | 28/375 | 22/399
Other Adverse Events (participants affected / at risk) | 163/375 | 176/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=375) | Ramipril (N=399)
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1
Myocardial infarction (Cardiac disorders) | 3 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Type III immune complex mediated reaction (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=375) | Ramipril (N=399)
Diarrhoea (Gastrointestinal disorders) | 28 | 24
Nausea (Gastrointestinal disorders) | 19 | 15
Oedema peripheral (General disorders) | 28 | 20
Nasopharyngitis (Infections and infestations) | 19 | 21
Upper respiratory tract infection (Infections and infestations) | 27 | 26
Urinary tract infection (Infections and infestations) | 21 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 22
Dizziness (Nervous system disorders) | 23 | 29
Headache (Nervous system disorders) | 41 | 54
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.